CLINICAL TRIAL: NCT00060021
Title: A Randomized, Placebo-Controlled, Blinded Study Of Acupuncture Therapy In Mucositis-Related Pain In Patients Undergoing Hematopoietic Stem Cell Transplantation
Brief Title: Acupuncture in Treating Mucositis-Related Pain Caused by Chemotherapy in Patients Undergoing Stem Cell Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Supportive Care
Other Study IDs: CDR0000299048; NCI-03-C-0125
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2004-04

CONDITIONS: Cancer
Keywords: oral complications; pain; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; chronic eosinophilic leukemia; primary myelofibrosis; chronic neutrophilic leukemia; chronic phase chronic myelogenous leukemia; de novo myelodysplastic syndromes; disseminated neuroblastoma; meningeal chronic myelogenous leukemia; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; ovarian choriocarcinoma; ovarian embryonal carcinoma; ovarian yolk sac tumor; ovarian immature teratoma; ovarian mature teratoma; ovarian monodermal and highly specialized teratoma; ovarian polyembryoma; ovarian mixed germ cell tumor; high risk metastatic gestational trophoblastic tumor; previously treated myelodysplastic syndromes; recurrent adult acute lymphoblastic leukemia; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent neuroblastoma; recurrent ovarian epithelial cancer; recurrent ovarian germ cell tumor; recurrent malignant testicular germ cell tumor; refractory chronic lymphocytic leukemia; relapsing chronic myelogenous leukemia; refractory hairy cell leukemia; refractory multiple myeloma; secondary acute myeloid leukemia; secondary myelodysplastic syndromes; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; stage II ovarian epithelial cancer; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult Burkitt lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III chronic lymphocytic leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III ovarian epithelial cancer; stage III malignant testicular germ cell tumor; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Burkitt lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV breast cancer; stage IV chronic lymphocytic leukemia; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV ovarian epithelial cancer; testicular choriocarcinoma and embryonal carcinoma; testicular choriocarcinoma and seminoma; testicular choriocarcinoma and teratoma; testicular choriocarcinoma and yolk sac tumor; testicular embryonal carcinoma and seminoma; testicular embryonal carcinoma and teratoma with seminoma; testicular embryonal carcinoma and teratoma; testicular embryonal carcinoma and yolk sac tumor with seminoma; testicular embryonal carcinoma and yolk sac tumor; testicular embryonal carcinoma; testicular teratoma; testicular yolk sac tumor and teratoma with seminoma; testicular yolk sac tumor and teratoma; testicular yolk sac tumor; recurrent adult acute myeloid leukemia; testicular choriocarcinoma; atypical chronic myeloid leukemia, BCR-ABL1 negative; myelodysplastic/myeloproliferative neoplasm, unclassifiable; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Neoplasms; Pain; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Neutrophilic, Chronic; Leukemia, Myeloid, Chronic-Phase; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Burkitt Lymphoma; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Neuroblastoma; Carcinoma, Ovarian Epithelial; Testicular Neoplasms; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Multiple Myeloma; Breast Neoplasms; Carcinoma, Embryonal; Seminoma; Teratoma; Endodermal Sinus Tumor; Teratoma, Testicular; Leukemia, Myeloid, Acute; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders; Lymphoma, B-Cell, Marginal Zone | interventions — Acupuncture Therapy; Analgesia

INTERVENTIONS:
Procedure: acupuncture therapy
Procedure: management of therapy complications
Procedure: pain therapy

SUMMARY:
RATIONALE: Acupuncture may be effective in relieving mucositis-related pain caused by chemotherapy in patients undergoing stem cell transplantation.

PURPOSE: Randomized clinical trial to study the effectiveness of acupuncture in treating mucositis-related pain caused by high-dose chemotherapy in patients who are undergoing stem cell transplantation.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of acupuncture vs placebo acupuncture in alleviating mucositis-related pain secondary to high-dose chemotherapy, as assessed by total cumulative dose of opioids used and subjective pain scores, in patients undergoing hematopoietic stem cell transplantation.
* Compare the overall number of patients requiring opioid therapy in these 2 intervention groups.
* Compare the nausea and vomiting scores of patients in these 2 intervention groups.
* Compare the sedation score of patients in these 2 intervention groups.
* Compare the use of other psychotropic medications (e.g., anxiolytics or hypnotics) in patients in these 2 intervention groups.
* Compare the need for total parenteral nutrition (TPN) and the number of days on TPN experienced by patients in these 2 intervention groups.
* Compare pruritus and the need for symptomatic treatment in patients in these 2 intervention groups.

OUTLINE: This is a randomized, double-blind, placebo-controlled study. Patients are stratified according to 9-phenylthiocarbamide/6-n-propylthiouracil (PROP) tasting ability (super-tasters vs non-super-tasters). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Beginning immediately after the development of mucositis pain, patients undergo acupuncture over 30 minutes once daily. Patients also receive standard pain management. Treatment continues until pain is completely resolved in the absence of unacceptable toxicity.
* Arm II: Patients undergo placebo acupuncture and receive standard pain management as in arm I.

PROJECTED ACCRUAL: A maximum of 45 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Must be undergoing hematopoietic stem cell transplantation (HSCT) through one of the following means:

  * Concurrent enrollment on a HSCT protocol with the Experimental Transplantation & Immunology Branch (ETIB) at the NCI Center for Clinical Research*
  * Receiving HSCT as a compassionate exemption following the clinical guidelines of an ETIB protocol*
* Directly observed oral or pharyngeal mucositis and/or suspected esophageal mucositis after high-dose chemotherapy
* No pain unrelated to mucositis requiring use of potent analgesics prior to initiation of high-dose chemotherapy NOTE: *Protocol must be known to generate more than 50% incidence of high-dose chemotherapy-induced mucositis

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* No history of bleeding disorders

Hepatic

* PT and PTT normal

Renal

* Not specified

Other

* No history or evidence of drug addiction or drug-seeking behavior
* No skin infection at the sites of acupuncture points

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No concurrent anticoagulant therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-03

CONTACTS AND LOCATIONS:
Overall Officials: Claude Sportes, MD, Study Chair — National Cancer Institute (NCI)
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States